CLINICAL TRIAL: NCT02224183
Title: Veterans Back to Health: A Study Comparing Yoga and Education for Veterans With Chronic Low Back Pain
Brief Title: Yoga vs. Education for Veterans With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Robert B Saper, BMC Attending Physician, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-32948; 3R01AT005956-05S1 (NIH)
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Recurrent Low Back Pain
Keywords: low back pain; yoga; education; Veterans; cost-effectiveness; military; back pain
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Educational Status; Yoga

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education (Active Comparator): Individuals randomized to the education group will receive The Back Pain Helpbook, an educational book with strategies for self-care including an exercise program, lifestyle modification, and tips for managing flare-ups. In addition, they will receive an assignment sheet outlining specific chapters to read over the course of the 12-weeks. In addition, participants receive at 3, 6, 9, and 12 weeks newsletters highlighting main points from the assigned chapters.
  Interventions: Behavioral: Education
- Yoga (Active Comparator): Weekly yoga classes will each be taught by two yoga instructors. Classes will be 75 minutes long. Mats and props will be provided. Yoga participants will be encouraged to practice for 30 minutes on days when they do not have class. They will be provided free of charge with a participant handbook, mat, block, and strap to aid home practice. Yoga home practice videos will be placed online for home practice and the website will track time spent using the videos for home practice. DVDs will be provided for those that do not have consistent access to the internet at home.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Education — Individuals randomized to the education group will receive The Back Pain Helpbook, an educational book with strategies for self-care including an exercise program, lifestyle modification, and tips for managing flare-ups. In addition, they will receive an assignment sheet outlining specific chapters to read over the course of the 12-weeks. In addition, participants receive at 3, 6, 9, and 12 weeks newsletters highlighting main points from the assigned chapters.
  Arms: Education
Behavioral: Yoga — Weekly yoga classes will each be taught by two yoga instructors. Classes will be 75 minutes long. Mats and props will be provided. Yoga participants will be encouraged to practice for 30 minutes on days when they do not have class. They will be provided free of charge with a participant handbook, mat, block, and strap to aid home practice. Yoga home practice videos will be placed online for home practice and the website will track time spent using the videos for home practice. DVDs will be provided for those that do not have consistent access to the internet at home.
  Arms: Yoga

SUMMARY:
Chronic low back pain (cLBP) is the most common pain condition in the military, causing substantial physical and psychological suffering, reduction in force readiness, and high economic cost. Yoga has been studied in 10 RCTs in civilian populations with cLBP suggesting it may be effective in reducing pain intensity, improving back-related function, and lowering pain medication use. Multiple differences exist between civilian and military populations with cLBP, making it necessary to adapt and test yoga for cLBP in military populations. This study's primary aim is to evaluate the effectiveness of yoga for reducing pain in military personnel and Veterans with cLBP through a structured, reproducible 12-week series of hatha yoga classes, supplemented with home practice, compared to an education group. Additionally, the enormous mental health burden often shouldered by returning military personnel presents another important distinguishing factor. Thus, the study's secondary aim is to assess yoga's capacity to reduce post-traumatic stress symptoms (PTSS). The third aim is to evaluate the cost-effectiveness of yoga for cLBP at 3 months and 6 months from the perspective of the provider, the Veteran, and the Veterans Health Administration. The fourth and final aim is to evaluate the effect of back pain and yoga on marital and family functioning. The proposed RCT will (1) establish a structured reproducible yoga protocol uniquely suited to Veterans populations with cLBP; (2) develop web-based delivery systems to assist Veterans in yoga home practice; (3) increase our knowledge of the feasibility and impact of yoga for Veterans' cLBP and psychological comorbidities. These results will help determine whether yoga is an effective modality for addressing cLBP in a Veteran population.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of any branch of military service
* Current low-back pain present for at least half the days over the past 6 months mean pain intensity for the previous week ≥4 on 0-10 rating scale

Exclusion Criteria:

* Significant yoga practice in the previous 6 months
* Have read The Back Pain Helpbook in the previous 6 months
* New LBP treatments started within the previous month or anticipated to begin in the next 3 months
* Known pregnancy
* Known inflammatory or systemic causes of LBP
* Severe and/or progressive medical, neurological, or psychiatric comorbidities
* Inability to understand/speak English
* Plans to move out of the area in the next 6 months
* Lack of informed consent
* Unwillingness to be randomized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in low back pain | Baseline, 6 weeks, 12 weeks, 24 weeks
  Measured using the Defense and Veterans Pain Rating Scale (DVPRS) which rates pain on a 0-10 scale
Change from baseline in back-related function | Baseline, 6 weeks, 12 weeks, 24 weeks
  Back-related function will be measured using the 23-point modified Roland Morris Disability Questionnaire (RMDQ).

SECONDARY OUTCOMES:
Change from baseline in pain medication use | Baseline, 6 weeks, 12 weeks, 24 weeks
  Pain medication use in the previous 7 days will be measured
Change from baseline in health-related quality of life | Baseline, 6 weeks, 12 weeks, 24 weeks
  Measured using the VR-12
Self-rated global improvement | 6 weeks, 12 weeks, 24 weeks
Patient satisfaction | Baseline, 6 weeks, 12 weeks, 24 weeks
  Measured using a single question that asks patients' overall satisfaction with their treatment
Change in post-traumatic stress symptoms | Baseline, 6 weeks, 12 weeks, 24 weeks
  Measured using PTSD Checklist - Civilian version (PCL-C)

OTHER OUTCOMES:
Change from baseline in post-concussive symptoms | Baseline, 12 weeks, 24 weeks
  Measured using the Neurobehavioral Symptom Inventory (NSI)
Change from baseline in sleep quality | Baseline, 12 weeks, 24 weeks
  Measured using the Pittsburgh Sleep Quality Index (PSQI)
Change from baseline in depressive symptoms | Baseline, 12 weeks, 24 weeks
  Measured using 9-item Patient Health Questionnaire (PHQ-9)
Change from baseline in anxiety symptoms (GAD-7) | Baseline, 12 weeks, 24 weeks
  Measured using the 7-item General Anxiety Disorder (GAD-7) questionnaire
Change from baseline in coping skills | Baseline, 12 weeks, 24 weeks
  Measured using the Coping Strategies Questionnaire (CSQ)
Change from baseline in self-efficacy | Baseline, 12 weeks, 24 weeks
  Measured using the Patient Self-Efficacy Questionnaire (PSEQ)
Marital/family functioning | Baseline, 12 weeks, 24 weeks
  Measured using the Dyadic Adjustment Scale (DAS)
Change in work status | Baseline, 12 weeks, 24 weeks
  Measured using the Work Productivity and Activity Impairment questionnaire
Cost-effectiveness | 6 weeks, 12 weeks, 24 weeks
  Medical record review and self-reported utilization data (medications, doctor visits, etc) will inform the cost effectiveness analysis of the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Saper, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Bedford VA Edith Nourse Rogers Memorial VA Hospital, Bedford, Massachusetts, United States

REFERENCES:
- [Derived] Roseen EJ, Pinheiro A, Lemaster CM, Plumb D, Wang S, Elwy AR, Streeter CC, Lynch S, Groessl E, Sherman KJ, Weinberg J, Saper RB. Yoga Versus Education for Veterans with Chronic Low Back Pain: a Randomized Controlled Trial. J Gen Intern Med. 2023 Jul;38(9):2113-2122. doi: 10.1007/s11606-023-08037-2. Epub 2023 Jan 17. PMID 36650329
- [Derived] Saper RB, Lemaster CM, Elwy AR, Paris R, Herman PM, Plumb DN, Sherman KJ, Groessl EJ, Lynch S, Wang S, Weinberg J. Yoga versus education for Veterans with chronic low back pain: study protocol for a randomized controlled trial. Trials. 2016 Apr 29;17(1):224. doi: 10.1186/s13063-016-1321-5. PMID 27129472